CLINICAL TRIAL: NCT05960253
Title: Comparison of the Peroperative Efficacy of Pericapsular Nerve Group Block and Lumbar Erector Spina Plan Block Applied Preoperatively in Patients Undergoing Hip Fracture Operation
Brief Title: Peroperative Effect of Regional Anesthesia in Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Levent Öztürk, Professor Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: hip surgery
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PENG block group (Active Comparator)
  Interventions: Procedure: Pericapsular Nerve Group Block
- L-ESP group (Experimental)
  Interventions: Procedure: Lumber Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block — 1st group to be applied PENG block
  Arms: PENG block group
Procedure: Lumber Erector Spinae Plane Block — 2nd group to be applied Lumber ESP block
  Arms: L-ESP group

SUMMARY:
A total of 120 patients scheduled for surgical operation due to hip fracture were divided into two randomized groups. The first group received pericapsular nerve group (PENG) block, while the second group received lumbar erector spinae plane (L-ESP) block prior to the surgery. Subsequently, all patients were positioned in the lateral decubitus position before spinal anesthesia and compared in terms of anesthesia effectiveness through pain scores.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists(ASA) 2-3 patients undergoing surgery due to hip fracture.

Exclusion Criteria:

* Patients in whom regional anesthesia is contraindicated.
* Patients who are unable to communicate.
* Patients with a known allergy to local anesthetics.
* Patients with organ failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Analgesia | 30 minutes
  Pain measurement via Visual Analog Scale (VAS) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)